CLINICAL TRIAL: NCT07118787
Title: Comparative Effects of Active Release Technique Verses Proprioceptive Neuromuscular Facilitation on Hamstring Flexibility in Patients Having Specific Low Back Pain
Brief Title: Active Release Technique Verses Proprioceptive Neuromuscular Facilitation on Hamstring Flexibility in Patients Having Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-/103-04/2022
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
Keywords: active release technique; low back pain; muscle stretching
MeSH Terms: conditions — Low Back Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: After screening the population based on inclusion and exclusion criteria, participants were included in the study. Participants signed a consent form regarding their willingness to participate in the study. The participants were divided equally into two groups where group one was evaluated for active release technique and group two was evaluated according to proprioceptive neuromuscular facilitation technique. The measurements were taken at baseline then at 2nd and at 4th week after the last Session. There were total 20 sessions, 5 sessions in a week for 4 weeks
Who Masked: Participant
Masking Description: The participants were randomly assigned in to two groups i.e. Group A and Group B by sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active release technique (Experimental): This group receives Active Release Technique applied on the hamstring muscle group to improve flexibility in patients with specific low back pain. Sessions are given at baseline then at 2nd and at 4th week after the last Session
  Interventions: Other: Active Release Technique
- Proprioceptive Neuromuscular Facilitation (Active Comparator): This group receives PNF stretching for the hamstring to enhance flexibility in patients with specific low back pain. Sessions are given at baseline then at 2nd and at 4th week after the last Session
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Active Release Technique — A manual therapy technique applied to release soft tissue tension in the hamstrings.
  Arms: active release technique
Other: Proprioceptive Neuromuscular Facilitation — A stretching technique involving passive stretching and isometric contractions of the hamstrings.
  Arms: Proprioceptive Neuromuscular Facilitation

SUMMARY:
The goal of this clinical trial is to learn whether Active Release Technique (ART) or Proprioceptive Neuromuscular Facilitation (PNF) is more effective in improving hamstring flexibility in adults with specific low back pain. It will also look at how these treatments affect pain and movement.

The main questions it aims to answer are:

Does ART or PNF improve hamstring flexibility more in people with specific low back pain?

Do participants report reduced pain and better movement after receiving either treatment?

Researchers will compare the effects of ART and PNF to see which method works better for improving flexibility and reducing pain.

Participants will:

Receive either ART or PNF therapy for 2 weeks

Attend regular physiotherapy sessions during the treatment period

Be assessed before and after treatment for hamstring flexibility and pain levels

DETAILED DESCRIPTION:
This randomized controlled trial was designed to compare the effectiveness of Active Release Technique (ART) and Proprioceptive Neuromuscular Facilitation (PNF) in improving hamstring flexibility among individuals with specific low back pain. Reduced hamstring flexibility is a common contributing factor in low back dysfunction, and identifying the most effective manual therapy technique can guide more targeted physical therapy interventions.

Participants were randomly assigned to receive either ART or PNF over a 2-week intervention period. Both groups received treatment administered by trained physiotherapists using standardized protocols. ART focused on applying specific manual pressure to soft tissues while moving the muscle through its range of motion, while PNF employed contract-relax stretching techniques to promote muscle lengthening and neuromuscular facilitation.

Participants were evaluated at baseline and after the completion of the intervention for changes in hamstring flexibility, with secondary observations on pain reduction and functional improvement. The study adhered to ethical standards, and all participants provided informed consent prior to participation.

The trial contributes to evidence-based physiotherapy by offering comparative insight into two widely used manual techniques in musculoskeletal rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having chronic low backache having hamstring tightness referred from orthopedic department
2. Patients having lumber disc budge, spinal spondylosis
3. Age group 25-40 years, having pain more than 3 months
4. Minimum 20-degree restriction in SLR unilaterally Both male and female

Exclusion Criteria:

1. Any history of injury in lower extremities in past 3 months
2. Knee osteoarthritis patients, knee deformities, discitis, osteomyelitis
3. Patients with injury of back, constant or severe persistent pain, inflammatory conditions (rheumatoid arthritis, ankylosing spondylitis, spinal infection lumber spondylolisthesis, and lumber spondylolysis.
4. Any pregnancy, history of previous surgery or fracture and history of radiculopathy or neuropathic pain.

   -

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Hamstring Flexibility (measured by Passive Straight Leg Raise Test) | at baseline then at 2nd and at 4th week after the last Session
  Flexibility of the hamstring muscle will be measured using a goniometer during the Passive Straight Leg Raise (SLR) test.

SECONDARY OUTCOMES:
Pain Intensity (measured by Numeric Pain Rating Scale - NPRS) | at baseline then at 2nd and at 4th week after the last Session
  Participants will rate their pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Montiha Azeem, DPT, Principal Investigator — University of Lahore
Locations (1):
- Lahore Poly Clinic, social security hospital, Lahore, Punjab Province, Pakistan